CLINICAL TRIAL: NCT03429062
Title: The Comparison of Community Based Personal Training to Whole Body Vibration on Balance and Gait Parameters in People With Multiple Sclerosis
Brief Title: Comparison of Two Community Based Exercise Protocols in People With Multiple Sclerosis
Status: Withdrawn | Type: Observational
Why Stopped: retirement of faculty PI
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Other Study IDs: 19517
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis
Keywords: balance; gait; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- personal training: Individuals with a diagnosis of MS and any level of function will be recruited to participate in exercise two times per week with trained personal trainers. Exercise consists of strengthening, stretching, balance, endurance and gait when able. Equipment to be used include treadmill, stationary bike, weight equipment.
  Interventions: Other: Personal training exercises
- Whole Body Platform: Individuals with a diagnosis of MS and able to walk with or without an assistive device will be recruited to participate in whole body platform training two times per week with a physical therapist. The exercise on the whole body platform includes strengthening, balance, stretching, and endurance for 30 second bouts. The whole body platform is on for 30 seconds then off. Each exercise will use the 30 seconds to complete.
  Interventions: Other: Personal training exercises

INTERVENTIONS:
Other: Personal training exercises — Personal training: strengthening, stretching, endurance, balance Whole body vibration: strengthening, balance, stretching, endurance, balance
  Other Names: whole body vibration platform exercise

SUMMARY:
This study will compare the benefits of two community based exercise programs, personal training and whole body vibration on balance and gait in people with Multiple Sclerosis. Anyone with a diagnosis of MS can participate in the personal training. Only people who can walk with or without an assistive device with a diagnosis of MS can participate in the Whole Body Vibration. Pre testing and post testing will be completed using balance and gait measures and self reporting measures for balance confidence and impact of MS. The program will run two times per week for six weeks.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a demyelinating disease of the central nervous system (CNS) that affects approximately 400,000 persons in the United States, and 1,200,000 persons between 16 and 65 years of age worldwide. It is a neurodegenerative pathology which can be characterized by a course of demyelination-mediated relapses and remissions, superimposed upon gradual neurologic deterioration, resulting in a clinical course that is unpredictable in its progression and severity. The pathophysiology associated with MS is the slowing or stopping of saltatory conduction of action potentials along myelinated axons in the CNS. This results in a clinical presentation that is varied and unpredictable in age of onset, disease progression, and the signs and symptoms experienced by each person with MS (PWMS).

Individuals with Multiple Sclerosis have a variety of symptoms before and after diagnosis. Common symptoms include double vision, partial loss of vision, numbness or weakness of the limbs, fatigue, depression, cognitive dysfunction, dizziness, tremor, decreased coordination, and unsteady gait. Many symptoms of MS are associated with increased fall risk similar to that found in older individuals.

The purpose of this study is to use and compare two different interventions in people with MS in a community setting. The first intervention is an assisted personal training program offered in a community setting to improve functional limitations and reduce risk for falls in people with MS. This exercise program will be provided by personal trainers educated in exercise training in people with MS. The personal training program is an ongoing program supported by the National MS Society. The second intervention is the use of Whole Body Vibration (WBV) platforms to improve gait ability and improve balance in people with MS.

Assisted personal training, circuit training has limited research in people with MS. This method of exercise is similar to exercise healthy individuals would complete in a fitness center setting with guidance from a personal trainer. In this study, the personal training program will be provided by educated personal trainers. These personal trainers completed a 24 hour continuing education course on exercise in people with neurodegenerative diseases. The facility, MindSet Charities has a strong ongoing personal training program for people with MS, and this program is supported by the National Multiple Sclerosis Society (NMSS). The individuals with MS attend 2 personal training sessions each week. The effectiveness of this type of program has not been studied to date.

There is a desire to improve training options to increase endurance, gait ability, and balance in people with MS. In the past decade whole body vibration has been studied in athletes, older individuals, people with chronic stroke, people with Parkinson Disease, and there are a few studies in people with MS. During WBV training, individuals stand on the platform and complete a series of exercises designed to improve gait ability and balance. The vertical vibrations during the session are thought to cause muscle contractions initiated by sensory receptors and reduce the recruitment threshold of motor units possibly resulting in increased activation of high threshold fast twitch muscle fibers.

Hypothesis:1. Individuals with MS who participate in either a personal training class or a WBV exercise protocol will have improvements in gait, balance, endurance, fatigue, and quality of life (QOL). 2. Individuals in the WBV training group will have a greater improvement in strength.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of MS,
* able to read, understand and sign the consent to participate form,
* adults between 18 and 85 years,
* attend a pre and post test session of 60-120 minutes

Exclusion Criteria:

* unable to read, understand the consent to participate form,
* unable to participate in any exercise

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes adults (18-85 years) with a diagnosis of Multiple Sclerosis. This is a sample of convenience, with recruitment occurring at MindSet Fitness and Yoga where exercise classes for people with MS occur every Tuesday and Thursday.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Mini Balance Evaluations Systems Test (MiniBEST Test) | 20 minutes
  Measure of dynamic balance, scores range from 0 (no Balance) to 28 good dynamic balance.

SECONDARY OUTCOMES:
Activities Specific Balance Scale | 15 minutes
  self report balance confidence, score from 0% (no confidence in balance) to 100% (full confidence in balance)
Fatigue Severity Scale | 10 minutes
  self report fatigue measure, scale goes from 1 (strongly agree with the statement about fatigue) to 7 (strongly disagree with statement about fatigue) higher score indicates less MS fatigue.
Multiple Sclerosis Impact Scale | 15 minutes
  Quality of life measure that measures the impact MS has on the persons day to day life. The scale ranges from 1 (not at all impactful) to 5 (extremely impactful), Scores range from 29 to 145. The higher the score the more they are impacted by MS in day to day life.
Dynamic Gait Index | 15 minutes
  Measure of gait, scale goes from 3 (normal) to 0 (unable) and range is 24 indicates normal gait, 0 indicates unable to walk, risk for falls is less than or equal to 19/24.
5 Times Sit to Stand Test | 1 minute
  Measure of strength and power, timed test, how long does it take to go from sit to stand, less than 15 secs is risk for falls.
2 Minute Walk test | 2 minutes
  measure of gait endurance, how far can the person walk in 2 minutes. Normal values 176-189 meters

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Csiza, PT, DSc, Principal Investigator — Texas Woman's University
Locations (1):
- MINDSET Fitness and Yoga, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No